CLINICAL TRIAL: NCT06702254
Title: Psychological Treatment Based on Cognitive Behavior Therapy Delivered by Mental Health Care Staff in Acute Psychiatric Inpatient Care.
Brief Title: Psychological Treatment in Psychiatric Inpatient Care.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Stockholm (Other Government)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Lena Reuterskiold, PhD, Region Stockholm
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-01169
Record Dates: First submitted 2024-11-08; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Anxiety and Depression; Psychiatric Inpatients
Keywords: Cognitive behavioral therapy; Acceptance and commitment therapy; Psychiatric inpatient care
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treament as usual (Other): The in-ward patient are provided treatment as usual. This can include medication, routine brief conversation and ward activity.
  Interventions: Other: Treatment as usual
- Psychological manualized treatment with CBT and ACT (Experimental): The intervention is based on a manual and is an add-on to treatment as usual. In-ward patients are offered a brief psychological treatment based on core features from CBT and ACT such as behavioral activation and work on values and unhelpful thoughts. Prior to the intervention nursing staff receive training in the manual followed by supervision during the treatment intervention. The treatment in this condition is an add-on to usual treatment given in the wards. The intervention is brief up to four sessions in the manual but can be shortened or extended to fit the patients admission time.
  Interventions: Behavioral: Experimental: Psychological manualized treatment with CBT and ACT

INTERVENTIONS:
Behavioral: Experimental: Psychological manualized treatment with CBT and ACT — The intervention is brief and centered around four therapeutic sessions that can be extended or shortened depending on how long patients are hospitalized. Core techniques from CBT and ACT are included in the manual and consists of behavioral activation and values and unhelpful thoughts. Nursing staff on these wards have received training in the manual parallel with supervision which is not given in the treatment as usual wards. The wards that have not received the intervention will be offered this at the end of their TAU period.
  Arms: Psychological manualized treatment with CBT and ACT
Other: Treatment as usual — This treatment as usual can consist of medication, brief talks, leisure activity on the wards.
  Arms: Treament as usual

SUMMARY:
There is a lack of psychological treatments within inpatient psychiatric care while there is support for active psychological interventions having an effect on psychiatric problems. The purpose of the present feasibility study is to test whether a psychological treatment based on Cognitive Behavioral therapy (CBT) and Acceptande and Commitment therapy (ACT) for patients in psychiatric inpatient care is acceptable, understandable, helpful and effective both for patients and the staff who carry out the treatment. The therapist in the project will receive training and on-going supervision in a CBT-manual created within the research group.

DETAILED DESCRIPTION:
The main questions the study aims to answer are:

1. Is cognitive behavioral therapy perceived as acceptable, comprehensible and helpful for patients in psychiatric inpatient ´care, when given by nursing staff in inpatient care?
2. Is cognitive behavioral therapy perceived as acceptable, understandable and helpful to the nursing staff who provided the treatment intervention?
3. Is cognitive behavioral therapy effective in reducing psychiatric symptoms such as depression, anxiety, and perceived health status for patients in psychiatric inpatient care when provided by nursing staff?

Participants are nursing staff from eight psychiatric inpatient wards and patients. The training consists of a two day workshop in the CBT manual followed by eight group supervision sessions parallell with patient treatment.

The patients are offered a CBT manual based psychological intervention with planned four treatment sessions but these can be flexibly prolonged to more sessions for repetition for patients staying for a longer period of time.

The study is a quasi-experimental design. Randomization takes place at ward level. The wards will be twin-matched based on patient problems and then randomized to treatment as usual (control group) or treatment as usual plus a CBT intervention (experimental group). Eight wards are included. Four wards will thus act as a control group and four wards as an experimental group. All within inpatient-care at Region Stockholm. The study aimed to include a total of 230 participants during 2020-2023. With a distribution ratio of 1:2, 77 participants are allocated to the experimental group and 153 participants to the control group, calculated on the basis of an expected effect size of 0.35 and a power of 0.8.

Patients who fulfill the inclusion criteria are informed about the study orally and in writing and are offered participation. Informed consent is collected upon offer of participation in the study. Patients are included consecutively as long as the ward and therapists have the available resources to accept more participants. Patients fill in self-report forms in connection with the usual enrollment and discharge routine. The self-report forms are questions about anxiety symptoms (GAD-7); perception of health (EQ-5D); depression symptoms (PHQ-9): experience of the intervention; Behavioral Activation Depression Scale-Short Form (BADS-SF); patient satisfaction. For the qualitative part with in-depth interviews, approx. 20 nursing staff are recruited. Semi-structured interview guide for nursing staff is created.

ELIGIBILITY:
Inclusion criteria:

* Meet criteria for and are enrolled in psychiatric inpatient care.
* Agree to participate in the study.
* Assessed to be stable enough to participate in a conversation after a routine ward medical assessment (do they understand what they are agreeing to/not to, can communicate, etc.)

Exclusion criteria:

* Other ongoing intensive psychotherapy (e.g. in outpatient care that continues during the psychiatric inpatient care stay).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-12-05 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Behavioral Activation Depression Scale-Short Form (BADS-SF) | Change from pre intervention to post intervention at treatment end, up to four weeks.
  A self-report with nine questions that measures current activity level and satisfaction linked to activity under the present week inclusive of today. Scale scores are from 0 to 6 with a maximum of 54. Higher scores indicate a greater level of activity and satisfaction.

SECONDARY OUTCOMES:
Generalized Anxiety Disorder-7 (GAD-7) | Change from pre intervention to post intervention at treatment end, up to four weeks.
  A self-report containing seven questions that measures various aspects of subjective worry, anxiety and stress over the course of the past two weeks. Minimum value is 0 and maximum value 3. Higher scores indicate more anxiety and worry.
Experience of Health (EQ-5D) (EuroQol, https://euroquol.org) | Change from pre intervention to post intervention at treatment end, up to four weeks.
  The EQ-5D is a self-report that consists of five dimensions: mobility, self care, daily activities, pain/discomfort, anxiety/depression. The EQ-5D also contains a visual analogue scale where patients can rate their overall health. Higher scores indicate better overall health and well being.
Patient Health Questionnaire (PHQ-9) | Change from pre intervention to post intervention at treatment end, up to four weeks.
  The PHQ-9 is a self-report with nine questions if patients have experienced depression, hopelessness or futility during the last two weeks. A minimum value of 0 and a maximum value of 3. Higher scores indicate more depression symtoms.
Patient Satisfaction (https://patientenkat.se/sv/) | Change from pre intervention to post intervention at treatment end, up to four weeks.
  A self-report used for all patients in psychiatric in-patient care nationally at discharge. The self-report contains five questions. Higher scores indicate more satisfaction with the in-patient care.
Experience of the psychological treatment | Post treatment, an average of two weeks.
  A self-report questionnaire created within the research group for this intervention. The self-report consists of seven questions that measures the patients experience of the intervention. The scores range from 1 to 7. Higher scores indicate a greater experience and satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Lena Reuterskiöld PhD, Principal Investigator — Region Stockholm
Locations (1):
- Psykiatri Nordväst, Stockholm, Sweden, Sweden

IPD SHARING:
Plan to Share IPD: No
IPD for this data set can not be made available on the individual participant level due to consent given by participants during project time since 2020. Although data on group level including measures of variance and details of statistical analysis plan will be shared to researchers on request.